CLINICAL TRIAL: NCT06610513
Title: Effect of Guided Imagery on Pregnancy Stress and Sleep Quality in Risky Pregnancy
Brief Title: Guided Imagery on Pregnancy Stress and Sleep Quality in Risky Pregnancy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Öznur Akçayüzlü, MsC, RN, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 126
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Effect of Guided Imagery Application on Pregnancy Stress and Sleep Quality in Risky Pregnant Women Will Be Checked
Keywords: Guided imagery; pregnancy; stress; sleep quality; risky pregnancy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Masking Description: Due to the study's nature, masking could not be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Guided imagery group (Experimental): Guided imagery will be applied to risky pregnant women in addition to normal nursing care.
  Interventions: Behavioral: Guided imagery
- control group (No Intervention): Only routine nursing care will be provided to risky pregnant women.

INTERVENTIONS:
Behavioral: Guided imagery — First meeting: The women will be introduced to the clinic, the purpose of the study will be explained, and a written consent form will be filled out. A Personal Information Form and the "Pregnancy Stress Assessment Scale" (GSDS-36) and the "Richard-Campbell Sleep Scale" will be filled out. After the questionnaires are filled out, the vital signs of the pregnant woman will be measured and then a 15-minute guided imagery video will be shown. The vital signs of the patient will be measured again 10 minutes after the guided imagery video is watched.
  Arms: Guided imagery group

SUMMARY:
In this thesis study, it is thought that with the guided imagery application to the hospitalized pregnant women, there will be a decrease in their stress levels and an increase in their sleep quality. In our country, there is no study where guided imagery application is used in risky pregnant women. It is thought that new information will be added to the literature as a result of this study. This study will be conducted to determine the effect of guided imagery application on pregnancy stress and sleep quality in risky pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Education level should be primary school or above
* Being in the 20th week of pregnancy or above
* Being planned to stay in the hospital for at least 5 days
* Being hospitalized for the first time during pregnancy
* Being within the first 3 days of hospitalization
* Knowing and speaking Turkish
* Being able to communicate verbally

Exclusion Criteria:

1. Having had guided imagery before
2. Having a diagnosis of mental illness
3. Having become pregnant through infertility treatment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women who have risky pregnancy will be included, therefore the study is gender based.
Enrollment: 48 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pregnancy Stress Assessment Scale | During 5 days after the first meeting with participant
  Pregnancy Stress Assessment Scale will be implemented to the pregnant women. The degree of anxiety, distress and worry experienced by pregnant women is "definitely not", "mild", "moderate", "serious" or "very serious" and is given on a score ranging from 0 to 4, and the perceived stress levels during pregnancy range from a minimum of 0 to a maximum of 144 points. As the score obtained from the scale increases, it is interpreted that stress increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Adana City Training and Research Hospital, Adana, Sariçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No